CLINICAL TRIAL: NCT04980612
Title: Feasibility Clinical Trial of Integrated Mind-Body Therapy for Chronic Low Back Pain
Brief Title: Development and Feasibility of Mindfulness Based Pain Reduction
Acronym: MBPR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: # 21-34357; 1R34AT010921 (NIH)
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low-back Pain
Keywords: pain; mindfullness; MBSR; Low Back; pain reduction; interoceptive awareness
MeSH Terms: conditions — Pain | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: The intervention and MBPR manual will be refined iteratively in 4 courses with 10 participants. The last of these 4 MBPR classes will be about 10 of 20 participants randomly assigned to either participate in standard MBSR or MBPR.
  The first part of the study is single-arm, the last randomized to assess acceptability of randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): 4 cohorts of 10 participants to MBPR (First 3 groups single-arm, final group of 10 randomly assigned to MBPR)
  Interventions: Behavioral: Mindfulness Based Pain Reduction
- Group 2 (Active Comparator): The last 20 participants will be randomly assigned to MBSR or MBPR, which will results in a control group with ~10 participants undergoing MBSR
  Interventions: Behavioral: Mindfulness Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness Based Pain Reduction — 40 participants will participate in a MBPR program. It will be an optimized mindfulness program specifically designed for treating cLBP that we will develop and test in this project. The format is the same as MBSR: 8 weeks of weekly 2½-hour group sessions and a daylong retreat.
  Arms: Group 1
Behavioral: Mindfulness Based Stress Reduction — 10 participants will participate in MBSR program. MBSR is a standardized and manualized 8-week program, delivered once a week in 2½-hour group sessions and a daylong retreat. It trains individuals in several mindfulness practices, e.g. focus on breath, varying degrees and directions of object orientation, open monitoring of awareness of intero- and exteroceptive stimuli and thoughts, de-reification (i.e. the notion that thoughts and perceptions are not always true to reality), and meta-awareness (i.e., awareness of thinking) in addition to focused attention.The program typically includes audio-recordings and a workbook for home practice and has shown benefits in patients with cLBP.
  Arms: Group 2

SUMMARY:
This is a development study with clinical outcomes. The investigators aim to develop and test an 8-week MBPR (Mindfulness-Based Pain Reduction) program, which draws on intervention work and clinical experience in the investigative team to optimize a mindfulness-based intervention for individuals with chronic pain. The overall goal of this study is to ensure that the MBPR program has been carefully refined and manualized in an in-person setting before performing clinical trials comparing MBPR to MBSR (Mindfulness-Based Stress Reduction) to test whether it improves pain outcomes.

This study includes a Pain Attention Task that separates insula activation during experimental heat application between different pain attention conditions.

DETAILED DESCRIPTION:
MBPR will be an optimized mindfulness program specifically designed for treating chronic low back pain (cLBP) that the investigators aim to develop and test in this project. 4 groups of 10 participants will receive MBPR consecutively to refine the MBPR curriculum. The format is the same as MBSR: 8 weeks of weekly 2½-hour group sessions and a daylong retreat. All sessions include training to enhance mindful interoceptive awareness through focused attention in the region of pain, the lower back.

A final group of 20 participants will be randomized to receive MBPR or MBSR. Total N=50 (40 MBPR; 10 MBSR). MBSR is a standardized and manualized 8-week program, delivered once a week in 2½-hour group sessions and a daylong retreat. It trains individuals in several mindfulness practices, e.g. focus on breath, varying degrees and directions of object orientation, open monitoring of awareness of intero- and exteroceptive stimuli and thoughts, de-reification (i.e. the notion that thoughts and perceptions are not always true to reality), and meta-awareness (i.e., awareness of thinking) in addition to focused attention. The program typically includes audio-recording and a workbook for home practice and has shown benefits in patients with cLBP.

This project also includes an ancillary brain imaging study designed to build on neuroscience reports of markedly decreased brain function and structure in the insular cortex (IC) of patients with cLBP. This project has the potential to reveal a potential central mechanism by which mind-body and acceptance-based approaches improve chronic pain conditions, e.g. cLBP. It may reveal a new paradigm for the treatment of cLBP with key importance and consequences for future behavioral intervention studies for pain.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic low back pain (cLBP) defined according to the NIH Research Task Force recommendation on Research Standards for cLBP: pain at least half the days in the past 6 months, by using 2 questions and a human figure drawing illustrating the region as the space between the lower posterior margin of the rib cage and the horizontal gluteal fold.
2. Average pain in the last month at least 3 out of 10 on Numeric Rating Scale [range 0 - 10, for 0 signifying no pain and 10 signifying worst pain imaginable]. This level of pain allows comparability of the study results with the majority of cLBP studies. Pain rated less than 3 is too mild to detect improvement.
3. Men and women aged 18 years old and older. The investigators are not enrolling younger children as they are not part of the Intensive Pain Rehabilitation Therapy program.
4. Eligibility will be assessed using the following questions: "(1) How long has back pain been an ongoing problem for you? and (2) How often has low-back pain been an ongoing problem for you over the past 6 months?" A response of greater than three months to question 1, and a response of "at least half the days in the past 6 months" to question 2 would meet the cLBP eligibility criterion.
5. Ability to speak English. We do not have the capacity, given the resources available in this proposal, to translate all course material and conduct groups into another language. The investiagtors have previously enrolled Hispanic participants into other studies who were fluent in English, and expect to do this in the proposed study.
6. Owning a smart phone

Exclusion Criteria:

1. Unable to provide informed consent.
2. A substance abuse, mental health, or medical condition that, in the opinion of investigators, will make it difficult for the potential participant to participate or that may need immediate changes in medical management that will affect study outcome measures. Such conditions may include cancer, liver failure, renal failure, pain conditions from inflammatory diseases (e.g. rheumatoid arthritis, ankylosing spondylitis, lupus), malignancies or abdominal aortic aneurysm, muscle weakness from radiculopathy. Radiculopathy or sciatic pain is NOT excluded as long as the condition is stable and does not lead to significant movement restrictions or <4/5 muscle weakness. Persons with significant substance abuse or mental health conditions that interfere with social functioning may be disruptive. Other medical or mental health conditions that need immediate changes in management need to be addressed before starting the study so that more reliable baseline measurements can be made. Patients who may need assessment for potentially necessary surgical interventions may not be able to complete the study. Regular opioid prescription is not an exclusion if stable over the past 3 months.
3. Spine related current or history of spine infection, spine tumor, vertebral fracture, cauda equina syndrome. Condition would increase heterogeneity of the sample.
4. Blindness, severe vision problems, deafness, severe hearing problems, bipolar or manic depression and not taking medication, major depression, psychoses (major), a substance abuse condition, dementia, unable to get up and down from the floor. Condition might make it difficult to participate.
5. Some other serious medical conditions that may alter key study outcomes, including untreated hypothyroidism, renal failure, and cirrhosis. Conditions that may alter key study outcomes.
6. Involvement in a lawsuit related to their back. Complicated medico-legal issues that could lead to individuals having a financial incentive to not report improvement.
7. Involved in Worker's Compensation claim.
8. Pregnant, breast-feeding, or planning to get pregnant in the next 12 months or less than 3 months post-partum. Particular back problems than may be associated with pregnancy and delivery may confound study outcomes.
9. Lack of stable housing or plan to move out of the area within the next 6 months.
10. MRI-related exclusion criteria: Cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), subjects who have ever been a metal worker/welder; history of eye surgery/eyes washed out because of metal, aortic aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, subjects with an I.U.D, a shunt (ventricular or spinal), electrodes, metal plates/ pins/screws/wires, or neuro/bio-stimulators (TENS unit), vision problems uncorrectable with lenses, claustrophobia; inability to lie still on one's back for approximately 60 minutes; prior neurosurgery; older tattoos with metal dyes; unwillingness to remove nose, ear or face jewelry, braces or permanent dental retainers. Iron-containing metal parts in the body can potentially be dislocated by strong magnetic fields and preclude assessment with MRI.
11. Received a steroid or botox injection in or near the spine in the last 3 months. This may alter key study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wolf E Mehling, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco; Osher Center for Intgerative Medicine, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MBPR: Mindfulness-Based Pain Reduction
- MBSR: Mindfulness-Based Stress Reduction
Period: Overall Study
Arm/Group | MBPR | MBSR
Started | 41 | 11
Completed | 34 | 6
Not Completed | 7 | 5
Not completed — Withdrawal by Subject | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MBPR | MBSR | Total
Number analyzed (Participants) | 41 | 11 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] — age in years
  years | 50.0 (12.1) | 58.4 (6.1) | 50.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 10 | 40
  Male | 11 | 1 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 36 | 11 | 47
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 9 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 26 | 6 | 32
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 0 | 2
PEG score [Mean (Standard Deviation); unit: units on a scale] — Pain, Enjoyment of Life and General Activity (PEG) combining Pain Intensity and Interference, 0 - 30 higher values indicate worse pain
  units on a scale | 14.2 (5.5) | 16.6 (4.9) | 14.8 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: Change in average pain intensity in past week on Numeric Rating Scale [0 to 10] will be assessed by internet-based questionnaire using REDCap negative values indicate improvement.
Time Frame: baseline, post 8-week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBPR | MBSR
Number analyzed (Participants) | 34 | 6
score on a scale | -2.30 (2.50) | -1.83 (1.94)

2. Secondary Outcome: Pain Interference
Description: Change in average of the scores for the 3 Pain Interference items on PROMIS-29 [5-point Likert scale from 1 "Not at all" to 5 "Very much"] average for past week will be assessed by internet-based questionnaire using REDCap [range 3 - 15, higher values more interference] negative numbers indicate improvement in pain interference
Time Frame: baseline, post 8-week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBPR | MBSR
Number analyzed (Participants) | 34 | 6
score on a scale | -6.23 (7.36) | -6.08 (3.22)

3. Other Pre Specified Outcome: Interoceptive Awareness
Description: change in scores for the 8 scales of the Multidimensional Assessment of Interoceptive Awareness (MAIA-2) [6-point 0-5 Likert scale Never to Always] will be assessed by internet-based questionnaire using REDCap. Each scale range from 0-5, total score over all 8 scales is the mean of the score of the 8 scales, also ranges 0-5. Higher values indicate higher interoceptive awareness.
  positive values indicate improvement.
Time Frame: baseline, post 8-week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBPR | MBSR
Number analyzed (Participants) | 34 | 6
score on a scale | 0.76 (0.61) | 0.61 (0.69)

4. Other Pre Specified Outcome: Changes in Insula Cortex Activation/Connectivity; Awaiting Separate Analysis
Description: using fMRI, insula cortex activation and connectivity in brain fMRI; awaiting separate analysis
Time Frame: baseline, post 8-week intervention.
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: 6 months
Description: minimal risk
Arm/Group | MBPR | MBSR
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/6
Other Adverse Events (participants affected / at risk) | 1/34 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBPR (N=34) | MBSR (N=6)
pain increase (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 — increased pain after a yoga movement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT04980612/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT04980612/SAP_001.pdf
  • Informed Consent Form (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT04980612/ICF_002.pdf